CLINICAL TRIAL: NCT06853106
Title: Digital-Based Multimodal Sleep Management Program for College Students with Insomnia: Randomized Controlled Trial
Brief Title: Digital Sleep Program for College Students with Insomnia
Acronym: DSP-CS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Pei-Shan, Tsai, Principal Investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202401041
Record Dates: First submitted 2025-02-20; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Insomnia
Keywords: Anxiety; Chronotypes; Daytime Sleepiness; Depression; Digital-based Sleep Management; Insomnia; Resilience; Sleep Reactivity; Mindfulness-based Breathing
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Disorders of Excessive Somnolence; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: We will implement a double-masking protocol, ensuring that assessors and data collectors are all blinded to group assignments. Additionally, group assignments will also be masked from the data analyzer to minimize potential bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Waitlist control group (Other): Participants in the waitlist control group will maintain their daily routines without receiving any intervention throughout the experiment.
  Interventions: Other: Waitlist control group
- digital-based multimodal sleep management program (Experimental): Participants in the experimental group will receive a 4-week digital-based multimodal sleep management program.
  Interventions: Behavioral: digital-based multimodal sleep management program

INTERVENTIONS:
Other: Waitlist control group — The participants in the waitlist control group will be informed that they are on a waiting list during the intervention period, serving as a no-treatment control. They will receive the sleep intervention (i.e., the digital-based sleep management program) four weeks after the intervention period is completed.
  Arms: Waitlist control group
Behavioral: digital-based multimodal sleep management program — The digital-based multimodal sleep management program consists of (1) sleep hygiene education, (2) sleep restriction, and (3) mindfulness breathing exercises. The program is internet-integrated and delivered via Google Meet, with 45-minute weekly sessions over four weeks. To increase participants' adherence to the sleep management program , the course instructor will request the participants to record their daily sleep diaries (time to bed, time to sleep, wake time during sleep and wake time) and sleep journals(practices of sleep hygiene, sleep restriction and mindfulness breathing exercise) in the mobile app for at least five consecutive days each week.
  Arms: digital-based multimodal sleep management program

SUMMARY:
This randomized controlled trial (RCT) study aims to evaluate the effectiveness of a digital-based multimodal sleep management program compared to a waitlist control group in improving sleep-related outcomes, including insomnia severity, daytime sleepiness, objective sleep parameters, and sleep reactivity to stress, as well as psychological health indices, such as depression, anxiety, and resilience. Additionally, this study seeks to examine the mediating role of different chronotypes in the effectiveness of the sleep intervention on the outcomes of interest.

DETAILED DESCRIPTION:
This is a parallel-group, randomized controlled trial (RCT). 90 participants who experiencing insomnia for at least 3 months with college students will be enrolled.

Eligible participants who complete the baseline measurements will be randomly allocated to a digital-based multimodal sleep management program group (N = 45) and a waitlist control group (N = 45).

The primary outcome is insomnia severity, assessed using the Insomnia Severity Index (ISI). The secondary outcomes include daytime sleepiness, objective sleep parameters, sleep reactivity, resilience, anxiety, and depression, which will be examined using the Epworth Sleepiness Scale (ESS), a wearable sleep tracker, the Ford Insomnia Response to Stress Test (FIRST), the Brief Resilience Scale (BRS), the State-Trait Anxiety Inventory (STAI), and the Beck Depression Index II (BDI-II), respectively. Additionally, chronotype will be assessed using the Morningness-Eveningness Questionnaire (MEQ) as a moderating role to be tested in this study. All outcomes will be measured at three time points: T0 (baseline assessment), T1 (immediately after the 4-week intervention period), and T2 (4 weeks after the intervention period).

ELIGIBILITY:
Inclusion Criteria:

1. Registered as a full-time student
2. Aged 18 to 26 years old
3. Experiencing insomnia for at least three months
4. Currently own and use a personal mobile device
5. Ability to read and speak Chinese
6. Not taking hypnotics, sedatives, or antidepressants
7. Not pregnant or lactating

Exclusion Criteria:

1. Using a smartphone model that cannot support the app
2. Currently using other sleep program apps
3. Meeting a STOP-BANG score of ≥3

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity:The Insomnia Severity Index (ISI) | T0 = baseline; T1 = immediately after intervention; T2 = 4 weeks after intervention.
  The Insomnia Severity Index (ISI) consists of seven items that assess the current perception of the severity of three insomnia symptoms. Each item is rated on a 5-point Likert scale, with the total score ranging from 0 to 28. Higher scores indicate greater severity of insomnia.

SECONDARY OUTCOMES:
Daytime Sleepiness:The Epworth Sleepiness Scale (ESS) | T0 = baseline; T1 = immediately after sleep intervention; T2 = 4 weeks after intervention.
  The Epworth Sleepiness Scale (ESS) is a self-reported measure of daytime sleepiness, assessing the propensity to doze or fall asleep during eight common daily activities. Each situation is rated on a 4-point scale, ranging from 0 ("would never doze") to 3 ("high chance of dozing"). The total score, obtained by summing the scores of the eight items, ranges from 0 to 24, with higher scores indicating greater levels of daytime sleepiness.
Sleep Parameters | T0 = baseline; T1 = immediately after sleep intervention; T2 = 4 weeks after intervention
  The sleep parameters will be recorded using a wearable sleep tracker (oCare Wrist-Worn Pro 100, Taiwan Biophotonic Corporation, Taiwan) daily for five consecutive days both before and immediately after the intervention. The wearable device will be paired with a mobile app for data collection and analysis. The sleep parameters derived from the device include sleep onset latency (SOL), wake after sleep onset (WASO), time in bed (TIB), total sleep time (TST), and sleep efficiency (SE).
Sleep Reactivity: The Chinese version of the Ford Insomnia Response to Stress Test (FIRST) | T0 = baseline; T1 = immediately after sleep intervention; T2 = 4 weeks after intervention
  The Ford Insomnia Response to Stress Test (FIRST) measures the extent to which sleep is affected by stress in individuals experiencing stressful conditions. It is a self-administered questionnaire consisting of nine questions, each rated on a 4-point scale, ranging from 1 (unlikely to happen) to 4 (very likely to happen). The total score ranges from 9 to 36, with higher scores indicating a greater degree of sleep disruption due to stress.
Resilience: The Chinese version of the Brief Resilience Scale (BRS) | T0 = baseline; T1 = immediately after sleep intervention; T2 = 4 weeks after intervention
  The Brief Resilience Scale (BRS) consists of six questions, each rated on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). Questions 1, 3, and 5 are forward-scored, while questions 2, 4, and 6 are reverse-scored. The total score ranges from 5 to 25, with higher scores indicating greater resilience, reflecting an individual's ability to adapt and recover from adverse events.
Depression: The Beck Depression Index II (BDI II) | T0 = baseline; T1 = immediately after sleep intervention; T2 = 4 weeks after intervention
  The Beck Depression Inventory-II (BDI-II) is a 21-item questionnaire designed to assess depressive symptoms. Response options range from 0 (did not feel it) to 3 (most or almost all the time). The total score ranges from 0 to 63, with higher scores indicating greater severity of depressive symptoms.
Anxiety: The State Trait Anxiety Inventory (STAI) | T0 = baseline; T1 = immediately after sleep intervention; T2 = 4 weeks after intervention
  The State-Trait Anxiety Inventory (STAI) is a self-report scale used to assess anxiety symptoms. It consists of 40 items, divided into two distinct dimensions: trait anxiety (20 items) and state anxiety (20 items). Each item is rated on a 4-point Likert scale, ranging from "almost never" to "almost always", with higher scores indicating greater levels of anxiety.

OTHER OUTCOMES:
Chronotype: The Chinese version of the Morningness-Eveningness Questionnaire (MEQ) | T0 = baseline; T1 = immediately after sleep intervention; T2 = 4 weeks after intervention
  The Morningness-Eveningness Questionnaire (MEQ) is a self-administered questionnaire consisting of 19 questions that assess an individual's preferred bedtime, wake-up time, and activity time. Responses are scored on a Likert-type scale, with total scores ranging from 16 to 86, reflecting differences in circadian rhythms. Higher scores indicate a stronger tendency to be a morning-type individual.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medicine University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No